CLINICAL TRIAL: NCT01486667
Title: Effect of Thyroxin Treatment in Sub Clinical Hypothyroidism Patients, on the Apnea Hypopnea Index Score, Lipid Profiles and Highly Sensitive CRP : A Randomized Double Blind Controlled Trial
Brief Title: Thyroxin Treatment in Sub Clinical Hypothyroidism, on the Apnea Hypopnea Index Score, Lipids and Highly Sensitive CRP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Anwar Ali Jammah, ASSISTANT PROFESSOR & CONSULTANT IN MEDICINE, ENDOCRINOLOGY, DIABETES & THYROID ONCOLOGY, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E-11-465
Record Dates: First submitted 2011-12-03; First posted 2011-12-06 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Dyslipidemia
Keywords: focus of study instead
MeSH Terms: conditions — Dyslipidemias | interventions — Thyroxine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sugar pill (Placebo Comparator)
  Interventions: Drug: sugar pill
- Levothyroxine (Active Comparator): Eligible patients will be randomized and be given 25 mcg of levothyroxine or identical placebo tablet at the beginning of the enrollment. The dosage of levothyroxine will subsequently be individualized for each patients. Serum levels of TSH and FT4 will be checked initially and then every 6 weeks until the end of the study. The investigators will attempt to maintain TSH levels between (0.25-2.5) mU/l which is the lower half of normal range. Advice given to patient regarding whether to increase or decrease the dose of medications will be based on patient TSH level according to study protocol.
  Interventions: Drug: levothyroxine

INTERVENTIONS:
Drug: levothyroxine — Eligible patients will be randomized and be given 25 mcg of levothyroxine or identical placebo tablet at the beginning of the enrollment. The dosage of levothyroxine will subsequently be individualized for each patients according to Serum levels of TSH and FT4 which will be checked initially and then every 6 weeks until the end of the study. The investigators will attempt to maintain TSH levels between (0.25-2.5) mU/l which is the lower half of normal range by adding or reducing the dose of levothyroxine. Advice given to patient regarding whether to increase or decrease the dose of medications will be based on patient TSH level according to study protocol.
  Arms: Levothyroxine
Drug: sugar pill — Eligible patients will be randomized and be given 25 mcg of levothyroxine or identical placebo tablet at the beginning of the enrollment. The dosage of drug will subsequently be individualized for each patients according to Serum levels of TSH and FT4 which will be checked initially and then every 6 weeks until the end of the study. The investigators will attempt to maintain TSH levels between (0.25-2.5) mU/l which is the lower half of normal range by adding or reducing the dose of medication. Advice given to patient regarding whether to increase or decrease the dose of medications will be based on patient TSH level according to study protocol.
  Arms: sugar pill

SUMMARY:
Obstructive sleep apnea (OSA) and hypothyroidism are both commonly found in clinical practice, and share a number of symptoms and clinical features. It has been shown that hypothyroid subjects are at high risk of developing sleep disorder breathing and OSA, and adequate thyroxine treatment may reduce the sleep disordered breathing.. However, the time-course and effect of treating subclinical hypothyroidism in OSA patients on the respiratory events during sleep is not known.

Subclinical hypothyroidism is associated with an increased risk of coronary heart disease (CHD). Dyslipidemia is a known complications of subclinical hypothyroidism and the effect of thyroxine treatment on lipid profile is controversial . Some reports suggested higher serum high-sensitivity C-reactive protein (hs-CRP), than healthy subjects; however, the effect of levothyroxine is controversial.

This project will help us to know if the treatment of subclinical hypothyroidism will improve the symptoms and reduce the progression of OSA, which may improve patients' quality of life by reducing the complication of OSA (hypertension, , depression, Cardiovascular diseases, etc.) or may even reduce mortality.It will help us to know the effect of subclinical hypothyroidism treatment on of lipid profiles and hs-CRP.

DETAILED DESCRIPTION:
Research Problem:

Obstructive sleep apnea (OSA) and hypothyroidism are both commonly found in clinical practice, and share a number of symptoms and clinical features. It has been shown that hypothyroid subjects are at high risk of developing sleep disorder breathing and OSA, and adequate thyroxine treatment may reduce the sleep disordered breathing.. However, the time-course and effect of treating subclinical hypothyroidism in OSA patients on the respiratory events during sleep is not known.

Subclinical hypothyroidism is associated with an increased risk of coronary heart disease (CHD). Dyslipidemia is a known complications of subclinical hypothyroidism (2)and the effect of thyroxine treatment on lipid profile is controversial . Some reports suggested higher serum high-sensitivity C-reactive protein (hs-CRP), than healthy subjects ; however, the effect of levothyroxine is controversial .

Research Significance:

This project will help us to know if the treatment of subclinical hypothyroidism will improve the symptoms and reduce the progression of OSA, which may improve patients' quality of life by reducing the complication of OSA (hypertension, , depression, Cardiovascular diseases, etc.) or may even reduce mortality.

It will help us to know the effect of subclinical hypothyroidism treatment on of lipid profiles and hs-CRP.

Research Objectives:

Primary objective:

• Effect of the treatment of subclinical hypothyroidism on the apnea hypopnea index (AHI) score.

Secondary objectives:

* Effect of the treatment of subclinical hypothyroidism on the lipid profile in patient with dyslipidemia.
* Effect of the treatment of subclinical hypothyroidism on hs-CRP

Research Methodology:

Patients with subclinical hypothyroidism will undergo first Polysomnography (PSG) (night 0) and laboratory investigations including lipid profiles and hc-CRP and then they will be enrolled and randomly assigned to receive either levothyroxine replacement therapy or identical placebo tablets in a blinded manner. The starting dose will be 25 mcg/day and the dose will be adjusted every 6 weeks to target TSH level between (0.25 -2.5 IU/mL). We will keep all patients on replacement dose for duration of 24 weeks. PSG will be performed twice only for OSA patient, after 12 weeks (night 1) and after 24 weeks (night 2). Lipid profile and hs-CRP will be done at the end of 24th weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old
* With Subclinical hypothyroidism defined as serum TSH concentration above 5.0 IU/mL when serum FT4 level is within the reference range
* With OSA defined as mild OSA: AHI 5 to 15/h; moderate OSA:AHI 15 to 30/h; and severe OSA: AHI greater than 30/h (30) will be enrolled.
* With confirmed sustained subclinical hypothyroidism, thus excluding patients with a temporary condition such as that in recovery from a non-thyroidal illness, measurement of TSH and FT4 will be conducted within four weeks before randomization.

Exclusion Criteria:

* Current treatment with Levothyroxine and lipid lowering medications or within two months before randomization.
* Conditions known to cause dyslipidemia e.g. uncontrolled diabetes mellitus (HbA1c >9), alcoholism and some medication use e.g. Estrogens. Glucocorticoids, Retinoids or Interferons.
* Conditions indicating levothyroxine treatment (34); including TSH levels more than 10 mU/l, clear symptoms or signs associated with thyroid failure and not related to OSA . e.g. goiter.
* State of pregnancy, Breast feeding or allergy to levothyroxine.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Effect of the treatment of subclinical hypothyroidism on the apnea hypopnea index (AHI) score. | 24 weeks

SECONDARY OUTCOMES:
Effect of the treatment of subclinical hypothyroidism on the lipid profile in patient with dyslipidemia and on hs-CRP | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University Sleep Disorders Center, Riyadh, Riyadh Region, Saudi Arabia